CLINICAL TRIAL: NCT06386107
Title: Association Between Thrombin Generation Parameters and the Risk of Bleeding in Patients Treated With Anticoagulants for Cancer Associated Thrombosis (CAT) (a Multicenter Study)
Brief Title: Thrombin Generation Parameters and Bleeding in Patients Treated With Anticoagulants for Cancer Associated Thrombosis
Acronym: CATforCAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Diagnostica Stago (Industry); LEO Pharma (Industry); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23PH188; 2023-A02175-40 (Other: ANSM)
Record Dates: First submitted 2024-01-22; First posted 2024-04-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Pulmonary Embolism; Thrombosis
Keywords: Cancer; Thrombosis; Anticoagulant associated bleeding
MeSH Terms: conditions — Neoplasms; Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Intervention Model Description: Prospective cohort of consecutive patients initiating full-dose anticoagulant therapy for an episode of CAT, followed up until the 6th month of treatment to assess the risk of clinically relevant adjunctive bleeding events and any other adverse event during anticoagulant therapy (recurrence of CAT, death).
  TGT measurement is fully automated and calibrated with quality control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with cancer associated thrombosis under curative anticoagulant treatment (Experimental): Patients with cancer associated thrombosis under curative anticoagulant treatment.
  Interventions: Biological: Thrombin Generation Assay (TGA)

INTERVENTIONS:
Biological: Thrombin Generation Assay (TGA) — Hemostasis is a complex process in which genetic or environmental conditions can cause shifts either towards pro-thrombotic states resulting in thrombosis, or towards pro-hemorrhagic states resulting in uncontrolled bleeding. Tests to assess a more global hemostatic profile, such as the TGA, have appeared as a more reliable alternative to assess the real hemostatic capacity of an individual. TGA is a global dynamic assay simultaneously and continuously measuring thrombin generation. It monitors the cleavage of a fluorigenic substrate that is simultaneously compared to the known thrombin activity in a non-clotting plasma sample.

SUMMARY:
Pulmonary embolism, the second leading cause of death in cancer patients, is effectively treated with anticoagulants. In patients with cancer-associated thrombosis (CAT), the use of anticoagulants is associated with 10 to 15% of bleeding in the first 6 months. Most of the guidelines propose to integrate the bleeding risk in the choice of therapies. Thrombin generation assay (TGA) reflects an overall hemostatic response and could be a useful biomarker. Proven on the thrombotic side in the CAT population, useful in the assessment of the bleeding risk of hemophiliac patients, the TGA is emerging as a tool. The investigators to measure TGA in cancer patients included prospectively, having recently developed a CAT and to evaluate the association between the measurement and the risk of hemorrhagic complication under anticoagulant during the first 6 month of treatment.

DETAILED DESCRIPTION:
Pulmonary embolism, the second leading cause of death in cancer patients, is effectively treated with anticoagulants. In patients with cancer-associated thrombosis (CAT), the use of anticoagulants is associated with 10 to 15% of bleeding in the first 6 months. Most of the guidelines propose to integrate the bleeding risk in the choice of therapies. Existing models for predicting anticoagulant associated bleeding risk applied to the CAT patients are not very predictive (AUC<0.60). Thrombin generation assay (TGA) reflects an overall hemostatic response and could be a useful biomarker. Proven on the thrombotic side in the CAT population, useful in the assessment of the bleeding risk of hemophiliac patients, the TGA is emerging as a tool. The investigators wish to measure TGA in cancer patients included prospectively, having recently developed a CAT and to evaluate the association between the measurement and the risk of hemorrhagic complication under anticoagulant during the first 6 month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active cancer, as defined by current French recommendations (Mahé I et al Rev Mal Respir 2021)
* Presenting acute proximal deep vein thrombosis of the lower limb (DVT) and/or proximal pulmonary embolism (at least segmental) (PE), confirmed by objective tests (Doppler ultrasound in the event of DVT; lung scintigraphy or CT scan in the event of PE)
* No contraindication for anticoagulant treatment at a curative dose at the time of inclusion

Exclusion Criteria:

* Patients participating in a therapeutic clinical trial with a blinded therapy or an open-label therapeutic trial who are included in the experimental treatment group.
* Patients already on anticoagulant at a curative dose for valvular or rhythmic embolic disease or a history of venous thromboembolic disease
* Hematological malignancies
* Patients with a contraindication to anticoagulant treatment on inclusion
* Patient whose relay by DOAC has already been carried out.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
The measurement of the area under the curve ( endogenious thrombin potential) nMxmin | during the first 6 months of treatment
  The measurment of the endogenious thrombin potential, during the first 6 months of treatment
the measurement of the lag time unit = seconds | during the first 6 months of treatment
  the measurement of the lag time, during the first 6 months of treatment
the measurement of the peak height unit = nm | during the first 6 months of treatment
  the measurement of the peak height during the first 6 months of treatment.
the measurement of the time to peak unit = seconds | during the first 6 months of treatment
  the mesearurement of the time to peak, during the first 6 months of treatment.

SECONDARY OUTCOMES:
Effect of adding TGT results on the performance of bleeding risk prediction scores | Month 1; Month 6
  Effect of adding TGT results on the performance (via AUC) of bleeding risk prediction scores.
Occurrence of clinically relevant bleeding between m1 and m6, based on the change in TGT | Month 1; Month 6
  Occurrence of clinically relevant bleeding between m1 and m6, based on the change in TGT (between inclusion and m1)
Occurrence of an event of interest under treatment | Month : 1 to 6
  Occurrence of an event of interest under treatment (recurrence of CAT, death, clinically relevant bleeding event) during the 6 months of follow-up, according to the TGT assessment at inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine POENOU, MD PHD, Principal Investigator — CHU SAINT-ETIENNE
Locations (4):
- France (4):
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - HCL, Lyon
  - Chu St-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No